# Effect of maxillary third molars extraction and non-extraction on distalization of first molars in a group of adolescent patients using infra-zygomatic gear distalizer

# A Randomized Clinical Trial

# **CONSENT FORM**

Submitted by

Nadeen Hafez Mohammed

Department of Orthodontics and Dentofacial Orthopedics.

Faculty of oral and dental medicine, future university in Egypt

**Date:** 15/8/2019



# RESEARCH ETHICS COMMITTEE Faculty of Oral and Dental Medicine (REC-FODM) CONSENT FORM

#### Title of Research

Effect of Maxillary Third Molar Extraction vs Non-extraction on Distalization of First molars in a Group of Adolescent patients Using Infra-Zygomatic Gear Distalizer:

A Randomized Clinical Trial

#### **Part I – Research Participant Information Sheet:**

- A. **Purpose of the Research**: is to compare the effect of the upper third molar presence and extraction on upper first molar infra-zygomatic mini-implant supported distalization.
- **B.** Description of the Research: this trial will assess the effect of third molar presence versus their extraction on distalization of maxillary first molars using infra-zygomatic mini-implant supported appliance to correct class II malocclusion.
- C. Potential Risks and Discomforts: pain associated with tooth movement, mini-implant insertion, and inflammation of mucosal tissues
- **D. Potential Benefits:** orthodontic treatment is done for the patient as indicated, improving patients' esthetics, function, and psychology by protrusion decrease.

| This Consent Document is approved for use by the Research Ethics Committee of FUE/FODM REC #: FUE.REC(14)/7-2019 | | _ |
|---|---|---|
| Date From: | To: | |



# Research Ethics Committees Faculty of Oral and Dental Medicine

- **E.** Cost: to participate in the research, you will bear no additional costs or extra loss.
- **F.** Compensation / Treatment: In the event of injury resulting from participation in this research study, Researcher will make a treatment to you, its facilities and professional attention. Financial compensation from FUE/FODM is not available.

#### **G. Voluntary Participation:**

Participation in this study is voluntary. You will suffer no penalty nor loss of any benefits to which you are otherwise entitled should you decide not to participate. Withdrawal from this research study will not affect your ability to receive alternative methods of Dental care available at FUE/FODM. Significant new findings developed during the course of the research study, which might be reasonably expected to affect your willingness to continue to participate in the research study will be provide to you.

#### H. Confidentiality:

C---4---4 D-----(-)

Your identity and medical record as a participant in this research study will remain confidential concerning any publications that may result from this study. Furthermore, your Dental/medical record may be reviewed by the Research Advisory Council or the agency sponsoring this research in accordance with applicable laws and regulations.

| $\overline{\mathbf{A}}$ | signed copy of the consent form will be given | to you |
|---|---|---|
| | | _ |
| I. | Contact Person(s): | |

| This Consent Document is approved for use by the | |
|------------------------------------------------------------------|-----|
| Research Ethics Committee of FUE/FODM REC # : FUE.REC(14)/7-2019 | |
| Date From: | To: |



#### PART II - Authorization for performance of certain procedures:

1. I/surrogate authorize **Dr. Nadeen Hafez Mohammed** and her associates to administer the following drugs, use the following devices or perform the following procedures during my treatment (or the treatment of the person named above for whom I am responsible)

**2.** I acknowledge that I have read, or had explained to me in a language I understand, the attached Research Participant Information sheet and that **Dr. Nadeen Hafez Mohammed** has explained to me the nature of the procedures described in the Research Participant Information Sheet as well as any benefits to be expected, possible alternative methods of treatment, the attendant discomforts and risks reasonably to be expected and the possibility that complications from both known and unknown causes may arise as a result thereof. I was given ample opportunity to comprehensively inquire about this study and procedures and all my questions were answered to my satisfaction.

- **3.** I understand that I am not entitled to reimbursement for expenses incurred as a result of my participation in this study
- **4.** I voluntarily accept the risks associated with the above-mentioned procedures with the knowledge and understanding that the extent to which they may be effective in my treatment (or the treatment of the patient named above, as the case may be) has not been established, that there may be side effects and complications from both known and unknown causes and that these procedures may not result in cure or improvement.
- 5. I understand that I am free to withdraw this consent and discontinue treatment with the above procedures at any time. The consequences and risks, if any, which might be involved in the event I later decide to discontinue such treatment have been

| This Consent Document is approved for use by the Research Ethics Committee of FUE/FODM REC # : FUE.REC(14)/7-2019 | |
|---|---|
| Date From: | To: |



### Research Ethics Committees Faculty of Oral and Dental Medicine

explained to me adequately. I understand that such withdrawal will not affect my ability to receive any dental/medical care made necessary by the performance of such studies or to which I might be otherwise entitled.

6. I confirm that I have read, or had read to me, the foregoing authorization and that all blanks or statements requiring completion were properly completed before I signed.

Patient Name:

| 1 attent Maine . | | | | |
|---|---|---|---|---|
| (If signed by Surrogate) | | | | |
| File #: | | | | |
| Patient/Surrogate: Signature | | | | |
| Relationship: | | | | |
| • | | _ | | |
| 7. I confirm that I have accurately translated ar | nd/or read the | information to the s | subject or his/her surrogat | Э. |
| Name: Nadeen Hafez Mohammed | | | | |
| Signature: | | | | |

**8.** I have fully explained to the above patient/ relative/ guardian the nature and purpose of the foregoing procedures, possible alternative methods of treatment which might be advantageous, the reasonable benefits to be expected, the attendant discomforts and risks involved, the possibility that complications may

This Consent Document is approved for use by the
Research Ethics Committee of FUE/FODM
REC # : FUE.REC(14)/7-2019

Date From:
To:

**FUE ID #: 20172999** 

Date:



# Research Ethics Committees Faculty of Oral and Dental Medicine

arise as a result thereof and the consequences and risks, if any, that might be involved in the event the patient/ relative/ guardian hereafter decides to discontinue such treatment.

It is my understanding that the above patient/ relative/ guardian understands the nature, purposes, benefits, and risks of participation in this research before signing this informed consent. I have also offered to answer any questions the above patient/ relative/ guardian might have with respect to such procedures and have fully and completely answered all such questions.

| ave fully and comp | etely answered all such questions | S. |
|---|---|---|
| Signature of Princ | pal Investigator/ Delegate): | |
| rint Name: Nade | n Hafez Mohammed | |
| Title: Master Stude | t at Future University in Egypt | |
| Oate: | | |
| This Consent Document is ap<br>Research Ethics Committee o | oved for use by the | |